CLINICAL TRIAL: NCT03370796
Title: Group Reminiscence Therapy for Elderly People With Cognitive Decline in Institutional Context
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: The Health Sciences Research Unit: Nursing (Unknown)
Responsible Party: Principal Investigator, Joao Apostolo, Professor Coordenador, Escola Superior de Enfermagem de Coimbra
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECOG_REM
Record Dates: First submitted 2017-11-30; First posted 2017-12-12 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Decline; Dementia; Cognitive Impairment
Keywords: dementia; cognitive impairment; cognition; quality of life; depressive symptoms; Reminiscence Therapy
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminiscence Therapy (Experimental): The Reminiscence program will consist of a set of sessions thematically sequenced topics that address the life course of the participant. Each session will integrate a group of activities that will be developed in group and will have a didactic character, privileging subjective interests and interpersonal communication.
  Interventions: Other: Reminiscence Therapy Program
- Control Group (No Intervention): The control group shall participate in the institutional care provided by the professionals of each RSE.

INTERVENTIONS:
Other: Reminiscence Therapy Program — The Reminiscence Therapy program is composed of: (i) main strand lasting 7 weeks, with sessions twice a week (total of 14 sessions); (ii) maintenance strand, which runs for 7 weeks, once a week (total of 7 sessions). The duration for each session will be 60 minutes.
  Arms: Reminiscence Therapy

SUMMARY:
The project presented here respond to this emerging need by implementing a Reminiscence Therapy program dedicated to elderly people in an institutional context. This will be a multicenter, randomized controlled study in which the participants' allocation will be made without their knowledge. Before the randomization process, the screening evaluation will be done, which will allow to verify the presence of the inclusion and exclusion criteria. The target population will be people age 65 or above years who present cognitive decline. After the randomization process, participants will be allocated randomly in the experimental group where the reminiscence program (composed by a main strand and maintenance strand) or in the usual institutional care group. The evaluation of the participants will be carried out individually and will take place in four different moments.This study will be conducted in RSE in the central region of Portugal.

DETAILED DESCRIPTION:
There are an estimated 46 million people with major Neurocognitive Disorders, and this figure is expected to increase to double every 20 years, with about 131.5 million people diagnosed by 2050 (Prince et al., 2015). The economic impact is significant, with costs estimated at US $ 818 million (Prince et al., 2015). In 2018, this value is expected to reach the trillion US dollar level, with serious implications for global societies and government authorities (Prince et al., 2015). Elderly people with cognitive decline progressively lose their cognitive capacities and experience motor disorders, leading, in more advanced stages of the disease, to family and carer burden, which often culminate in their institutionalization.

According to Kuske et al. (2009), about 60% of all institutionalized people in industrialized countries present some form of dementia, which poses new challenges for these institutions and for its professionals. This process is inevitably associated with an increase in the prevalence of chronic degenerative diseases, particularly neurocognitive disorders (NCD). The category of NCD includes all the disorders in which the primary clinical deficit is in cognitive function, being this deficit acquired (documented by standardized neurological tests or by quantitative clinical evaluation), that is, it represents a decline from a previous functional level (APA, 2013).

In this sequential line, priority is given to the design of interventions that effectively focus on the stimulation of best practices for active aging, aiming at the implementation of measures that minimize the impact of NCD by slowing down their progression or modulating their associated symptomatology (Directorate General for Health, 2016). Knowing that the drugs introduced so far in clinical practice are restricted to symptomatic control, not being able to prevent the progression of the disease, non-pharmacological interventions have been gaining special prominence. The literature emphasizes the value of Reminiscence as a strategy for people with cognitive deficits. This stimulating intervention is based on the recovery of significant life events with special focus on resolving past conflicts.

Reminiscence is a pleasant and stimulating activity that contributes to the reduction of social isolation, revealing itself as a strategy to promote interpersonal relations (Cooney et al., 2014; Gibson, 2004). It has been reported as an intervention associated with pleasure, safety and sense of belonging (Cappeliez & O'Rourke, 2006). It is also a low-cost therapeutic option (Siverová & Bužgová, 2014). In addition, according to Westerhof, Bohlmeijer and Webster (2010), the exchange of autobiographical memories through Reminiscence, even in the final stages of the dementia, can produce considerable and measurable gains that are reflected in increased levels of well-being, decreased depression levels and improved cognitive function as well as increased verbal fluency.

In view of the above, it is considered that the implementation of a structured Reminiscence program can maximize cognitive functioning, improve depressive symptoms and promote quality of life by facilitating the adaptation process and contributing to the promotion of the dignity of people with cognitive decline and who are in Day Care regime or living in Residential Structures for the Elderly (RSE).

ELIGIBILITY:
Inclusion Criteria:

* have the capacity to informally consent participation in the study;
* have the ability to remain in a group within 60 minutes;
* have sufficient auditory capacity to participate in discussions;
* have sufficient visual capacity to see the materials that are part of the applied program;
* have criteria of cognitive decline.

Exclusion Criteria:

* present an unstable clinical condition;
* do not wish to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the participant's Cognition | Intermediate assessment (week 7)
  Outcome Measure - Montreal Cognitive Assessment (MoCA)
Change from Baseline in the participant's Cognition | Post-intervention assessment (week 14)
  Outcome Measure - Montreal Cognitive Assessment (MoCA)
Change from Baseline in the participant's Cognition | Five-week follow-up assessment (week 19)
  Outcome Measure - Montreal Cognitive Assessment (MoCA)
Change from Baseline in the participant's Depressive Symptoms | Intermediate assessment (week 7)
  Outcome Measure - Geriatric Depression Scale - 10 itens version (GDS-10)
Change from Baseline in the participant's Depressive Symptoms | Post-intervention assessment (week 14)
  Outcome Measure - Geriatric Depression Scale - 10 itens version (GDS-10)
Change from Baseline in the participant's Depressive Symptoms | Five-week follow-up assessment (week 19)
  Outcome Measure - Geriatric Depression Scale - 10 itens version (GDS-10)
Change from Baseline in the participant's Quality of Life | Intermediate assessment (week 7)
  Outcome Measure -World Health Organization Quality of Life-Older Adults Module (WHOQOL-OLD)
Change from Baseline in the participant's Quality of Life | Post-intervention assessment (week 14)
  Outcome Measure -World Health Organization Quality of Life-Older Adults Module (WHOQOL-OLD)
Change from Baseline in the participant's Quality of Life | Five-week follow-up assessment (week 19)
  Outcome Measure -World Health Organization Quality of Life-Older Adults Module (WHOQOL-OLD)

CONTACTS AND LOCATIONS:
Overall Officials: João LA Apóstolo, PhD, Principal Investigator — Nursing School of Coimbra
Locations (1):
- Health Sciences Research Unit: Nursing, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuske B, Luck T, Hanns S, Matschinger H, Angermeyer MC, Behrens J, Riedel-Heller SG. Training in dementia care: a cluster-randomized controlled trial of a training program for nursing home staff in Germany. Int Psychogeriatr. 2009 Apr;21(2):295-308. doi: 10.1017/S1041610208008387. Epub 2009 Feb 5. PMID 19193252
- [Background] Directorate-General for Health. (2016). Portugal Saúde Mental em Números - 2015. Programa Nacional para a Saúde Mental. 75-86. Retrieved from http://www.apah.pt/media/publicacoes_tecnicas_sector_saude_2/Saude_Mental.pdf
- [Background] APA (213). Diagnostic and statistical manual of mental disorders (5th ed).(American Psychiatric Association, Ed.). Arlington.
- [Background] Cooney A, Hunter A, Murphy K, Casey D, Devane D, Smyth S, Dempsey L, Murphy E, Jordan F, O'Shea E. 'Seeing me through my memories': a grounded theory study on using reminiscence with people with dementia living in long-term care. J Clin Nurs. 2014 Dec;23(23-24):3564-74. doi: 10.1111/jocn.12645. Epub 2014 Jul 12. PMID 25040857
- [Background] Gibson, F. (2004). The past in the present: Using reminisce in health and social care. Baltimore: Health Professions Press.
- [Background] Cappeliez P, O'Rourke N. Empirical validation of a model of reminiscence and health in later life. J Gerontol B Psychol Sci Soc Sci. 2006 Jul;61(4):P237-44. doi: 10.1093/geronb/61.4.p237. PMID 16855036
- [Background] Siverová, J., & Bužgová, R. (2014). Influence Reminiscence Therapy on Quality of Life Patients in the Long-Term Hospital. Central European Journal of Nursing and Midwifery, 5 (1), 21-28
- [Background] Westerhof, G. J., Bohlmeijer, E., & Webster, J. D. (2010). Reminiscence and mental health: A review of recent progress in theory, research and interventions. Ageing and Society, 30 (04), 697-721.
- [Background] Prince, M., Wimo, A., Guerchet, M., Ali, G., Wu, Y., & Prina, M. (2015). World Alzheimer Report 2015 The Global Impact of Dementia. Alzheimer's Disease International. Retrieved from https://www.alz.co.uk/research/WorldAlzheimerReport2015.pdf